CLINICAL TRIAL: NCT04382963
Title: Stroke Prevention in the Wisconsin Native American Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1550; A535700 (Other: UW Madison); SMPH/NEURO SURG/NEURO SURG (Other: UW Madison); Protocol Version 11/12/2020 (Other: UW Madison)
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Atherosclerosis
Keywords: Stroke; Atherosclerosis; Native American; Risk factor modification; Proteonomics; Genomics
MeSH Terms: conditions — Stroke; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Risk- intense coaching (Other): age ≥ 55 with MORE than three of the following risk factors:
  * History of TIA/Stroke
  * History of Coronary Artery disease
  * History of Hypertension and/or current elevated blood pressure
  * History of Diabetes
  * Current smoker
  * BMI ≥30
  Interventions: Other: High Risk - intensive coaching
- High Risk - standard care (Other): age ≥ 55 with MORE than three of the following risk factors:
  * History of TIA/Stroke
  * History of Coronary Artery disease
  * History of Hypertension and/or current elevated blood pressure
  * History of Diabetes
  * Current smoker
  * BMI ≥30
  Interventions: Other: High Risk - standard care
- Low risk - control (Other): age ≥ 55 with LESS than three of the following risk factors:
  * History of TIA/Stroke
  * History of Coronary Artery disease
  * History of Hypertension and/or current elevated blood pressure
  * History of Diabetes
  * Current smoker
  * BMI ≥30
  Interventions: Other: Low Risk - control

INTERVENTIONS:
Other: High Risk - intensive coaching — The following assessment will occur: health assessment, blood pressure, BMI, history TIA/stroke, blood mRNA and protein analysis, ultrasound, cognitive assessment, stroke education, intensive coaching face-to-face.
  Furthermore, this group will receive intensive initiation of the American Heart Association Guidelines for Management of Risk Factors with individual face-to-face coaching meetings on lifestyle change and adherence to treatment on at a least quarterly basis.
  Arms: High Risk- intense coaching
Other: High Risk - standard care — The following assessment will occur: health assessment, blood pressure, BMI, history TIA/stroke, blood mRNA and protein analysis, ultrasound, cognitive assessment, stroke education.
  Arms: High Risk - standard care
Other: Low Risk - control — Control participants will undergo the same study events as the Low Risk group, except without receiving information and advice about eliminating stroke risk factors.
  Arms: Low risk - control

SUMMARY:
This project will develop a "Stroke Awareness Team" including training of Oneida Health Service Coaches working in partnership with the UW team for a population-based health awareness program. This team will develop a series of Oneida Nation Healthy Living and Stroke Awareness Events (from now on health events) to provide education as to the severity of the problem as well as our standard therapies for lifestyle change and risk factor avoidance. This will include education of the healthy members of the tribe including the children to identify signs of stroke and TIA in their elders as well as to develop healthy lifestyles at the earliest of ages to influence the elders to modify their risks.

DETAILED DESCRIPTION:
The study will enroll 100 high risk tribe members and 20 low stroke risk tribe members. Each of these will be further studied for their atherosclerotic load by ultrasound measurements at the carotid bifurcation for presence of plaque as well as its stability or instability during pulsation. Enrolled participants will also receive assessment of biomarkers for stroke risk, including stroke-related vascular cognitive decline, an early and modifiable marker of TIA risk and serum analysis for glucose, cholesterol, microRNA and key proteins felt to be biomarkers of stroke.

The high risk participants will be randomized into two groups, and data analyzed by gender, age, history of cerebrovascular events, and the presence or absence of atherosclerosis in their carotid bifurcation including equal numbers of participants that in spite of high risk, have not yet deposited plaque.

* One group will receive advice about standard therapy and information concerning risk factor guidelines to improve health awareness.
* The other group will receive the same plus intensive initiation of the American Heart Association Guidelines for Management of Risk Factors with at least quarterly individual face-to-face coaching meetings on lifestyle change and adherence to treatment.

At the end of 2-year follow-up, all groups will be reassessed for adherence to the program, atherosclerotic plaque progression or regression and its stability, serum biomarker response to therapy interventions, successful risk factor modification, vascular cognitive decline and incidence of stroke and TIA. Intention to treat analysis will estimate the efficacy of health coaching and will use G-estimation to correct for issues of non-compliance and discontinuation. Groups will be compared for change in both risk factors and outcomes.

Vascular cognitive decline is an important symptom of cerebrovascular disease which may precede a physical stroke with devastating results. Extensive preliminary data show that the frequency of this is surprisingly common in high risk patients and may predispose patients to later dementia. Vascular cognitive decline is a risk factor for stroke, but also is modifiable. A prior small study showed that intervention could stop the rate of decline. The study will see if this predicts participants at greatest risk for stroke that would improve with an intensive intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving health care through the Oneida Health Council Program
* Participants deemed to be at high risk for stroke by modified Framingham assessment of medical history, including cerebral cardiovascular symptomatology, hypertension, diabetes, smoking, BMI
* Willingness to participate in the study, including two-year follow-up
* Controls will be selected using the same criteria with the exception that upon screening, they are not deemed to be at high risk for stroke.

Exclusion Criteria:

* Presence of established dementia
* Inability to participate in physical and exercise programs due to preexisting disability
* Illiteracy
* Prior carotid procedure altering ultrasound finding
* Presence of medical condition precluding participation or follow-up over a two-year period of time.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Incidence of Stroke or TIA | baseline and 2 years
  Number of incidences of stroke or TIA during the study
Change in Number of Participants that meet AHA Simple Rules for Diastolic Blood Pressure | baseline and 2 years
  Number of Participants with diastolic blood pressure < 90 mmHg
Change in Number of Participants that meet AHA Simple Rules for Systolic Blood Pressure | baseline and 2 years
  Number of Participants with systolic blood pressure < 140 mmHg
Change in Number of Participants that meet AHA Simple Rules for Total Cholesterol | baseline and 2 years
  Number of Participants with total cholesterol < 200 mg/dL
Change in Number of Participants that meet AHA Simple Rules for Low Density Lipoprotein Cholesterol (LDL-C) | baseline and 2 years
  Number of Participants with LDL-C < 100 mg/dL
Change in Number of Participants that meet AHA Simple Rules for High Density Lipoprotein Cholesterol (HDL-C) | baseline and 2 years
  Number of Participants with HDL-C > 60 mg/dL
Change in Number of Participants that meet AHA Simple Rules for Blood Sugar | Baseline and 2 years
  Number of Participants with A1c < 7.5
Change in Number of Participants that meet AHA Simple Rules for Body Mass Index (BMI) | Baseline and 2 years
  Number of Participants who improve BMI
Change in Number of Participants that meet AHA Simple Rules for Smoking Status | baseline and 2 years
  Number of Participants who Smoke
Change in TabCAT Score | baseline and 2 years
  The Tablet-based Cognitive Assessment Tool will examine avorites (rote verbal learning and memory), match (processing speed), flanker (executive functions), and line orientation (visuospatial abilities).
Change in Montreal Cognitive Assessment (MoCA) Vancouver Island Coastal First score | baseline and 2 years
  Montreal Cognitive Assessment will assess vascular cognitive decline

SECONDARY OUTCOMES:
Change in Plaque Area | baseline and 2 years
  Measured via carotid ultrasound.
Change in pulsatility index in carotid arteries | baseline and 2 years
  Measured via carotid ultrasound. This index is a unitless measurement calculated: peak systolic velocity - end diastolic velocity, divided by the mean velocity, higher values are thought to represent increased resistance to blood flow
Correlation of carotid plaque grayscale texture features (grayscale median values [no units]) to stroke risk factors | baseline and 2 years
  Measured via carotid ultrasound
Change in Circulating Dipeptidyl Peptidase (DPPIV) | Baseline and 2 years
  DPPIV is a circulating protein associated with cardiovascular risk. This will be measured via blood draw at baseline and 2 years.
Change in Circulating Galectin3 (Gal-3) | baseline and 2 years
  Gal-3 is a circulating protein associated with cardiovascular risk. This will be measured via blood draw at baseline and 2 years.

OTHER OUTCOMES:
Change in Serum microRNA | baseline and 2 years
  Levels of serum microRNA are associated with increased stroke risk. This will be measured via blood draw at baseline and 2 years.
Compliance Rates | 2 years
  Number of people complying with study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dempsey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Oneida Comprehensive Health Division, Oneida, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Following transparency and reproducibility guidelines (NIH NOT-OD-15-103), the data resulting from this research proposal will be made publicly available. This will help ensure that other researchers are able to reproduce and/or extend our findings, and will enhance the scientific rigor of this proposal. Data will be made available for download to any individual or organization who requests data and abides by a data-sharing agreement that will be developed. This agreement will require that the data be used solely for research, that individuals or organizations secure the data using conventional electronic safeguards, and that once data analysis is complete, the data be destroyed. In general, data acquired in this study will be made available publicly after initial key manuscripts have been accepted for publication. Manuscripts will include relevant methodological details to allow for reproducibility by other researchers and the ability to extend or findings.

REFERENCES:
- [Background] Harris R, Nelson LA, Muller C, Buchwald D. Stroke in American Indians and Alaska Natives: A Systematic Review. Am J Public Health. 2015 Aug;105(8):e16-26. doi: 10.2105/AJPH.2015.302698. Epub 2015 Jun 11. PMID 26066955
- [Background] Berman SE, Wang X, Mitchell CC, Kundu B, Jackson DC, Wilbrand SM, Varghese T, Hermann BP, Rowley HA, Johnson SC, Dempsey RJ. The relationship between carotid artery plaque stability and white matter ischemic injury. Neuroimage Clin. 2015 Aug 22;9:216-22. doi: 10.1016/j.nicl.2015.08.011. eCollection 2015. PMID 26448914
- [Background] Darwish MA, Hammon WM. Studies on Japanese B encephalitis virus vaccines from tissue culture. VI. Development of a hamster kidney tissue culture inactivated vaccine for man. 3. Potency testing of an attenuated strain of OCT-541. J Immunol. 1966 May;96(5):878-84. No abstract available. PMID 4288023
- [Background] Wesley UV, Hatcher JF, Ayvaci ER, Klemp A, Dempsey RJ. Regulation of Dipeptidyl Peptidase IV in the Post-stroke Rat Brain and In Vitro Ischemia: Implications for Chemokine-Mediated Neural Progenitor Cell Migration and Angiogenesis. Mol Neurobiol. 2017 Sep;54(7):4973-4985. doi: 10.1007/s12035-016-0039-4. Epub 2016 Aug 15. PMID 27525674
- [Background] Amersfoort J, Schaftenaar FH, Douna H, van Santbrink PJ, Kroner MJ, van Puijvelde GHM, Quax PHA, Kuiper J, Bot I. Lipocalin-2 contributes to experimental atherosclerosis in a stage-dependent manner. Atherosclerosis. 2018 Aug;275:214-224. doi: 10.1016/j.atherosclerosis.2018.06.015. Epub 2018 Jun 13. PMID 29960897
- [Background] Hochmeister S, Engel O, Adzemovic MZ, Pekar T, Kendlbacher P, Zeitelhofer M, Haindl M, Meisel A, Fazekas F, Seifert-Held T. Lipocalin-2 as an Infection-Related Biomarker to Predict Clinical Outcome in Ischemic Stroke. PLoS One. 2016 May 6;11(5):e0154797. doi: 10.1371/journal.pone.0154797. eCollection 2016. PMID 27152948
- [Background] Greenland S, Lanes S, Jara M. Estimating effects from randomized trials with discontinuations: the need for intent-to-treat design and G-estimation. Clin Trials. 2008;5(1):5-13. doi: 10.1177/1740774507087703. PMID 18283074
- [Background] Vermeer SE, Prins ND, den Heijer T, Hofman A, Koudstaal PJ, Breteler MM. Silent brain infarcts and the risk of dementia and cognitive decline. N Engl J Med. 2003 Mar 27;348(13):1215-22. doi: 10.1056/NEJMoa022066. PMID 12660385
- [Background] Tyas SL, Salazar JC, Snowdon DA, Desrosiers MF, Riley KP, Mendiondo MS, Kryscio RJ. Transitions to mild cognitive impairments, dementia, and death: findings from the Nun Study. Am J Epidemiol. 2007 Jun 1;165(11):1231-8. doi: 10.1093/aje/kwm085. Epub 2007 Apr 12. PMID 17431012
- [Background] Mitchell CC, Stein JH, Cook TD, Salamat S, Wang X, Varghese T, Jackson DC, Sandoval Garcia C, Wilbrand SM, Dempsey RJ. Histopathologic Validation of Grayscale Carotid Plaque Characteristics Related to Plaque Vulnerability. Ultrasound Med Biol. 2017 Jan;43(1):129-137. doi: 10.1016/j.ultrasmedbio.2016.08.011. Epub 2016 Oct 5. PMID 27720278
- [Background] Jackson DC, Sandoval-Garcia C, Rocque BG, Wilbrand SM, Mitchell CC, Hermann BP, Dempsey RJ. Cognitive Deficits in Symptomatic and Asymptomatic Carotid Endarterectomy Surgical Candidates. Arch Clin Neuropsychol. 2016 Feb;31(1):1-7. doi: 10.1093/arclin/acv082. Epub 2015 Dec 10. PMID 26663810
- [Background] Dempsey RJ, Jackson DC, Wilbrand SM, Mitchell CC, Berman SE, Johnson SC, Meshram NH, Varghese T, Hermann BP. The Preservation of Cognition 1 Year After Carotid Endarterectomy in Patients With Prior Cognitive Decline. Neurosurgery. 2018 Mar 1;82(3):322-328. doi: 10.1093/neuros/nyx173. PMID 28575478
- [Background] Dempsey RJ, Varghese T, Jackson DC, Wang X, Meshram NH, Mitchell CC, Hermann BP, Johnson SC, Berman SE, Wilbrand SM. Carotid atherosclerotic plaque instability and cognition determined by ultrasound-measured plaque strain in asymptomatic patients with significant stenosis. J Neurosurg. 2018 Jan;128(1):111-119. doi: 10.3171/2016.10.JNS161299. Epub 2017 Mar 10. PMID 28298048
- [Background] Mitchell CC, Wilbrand SM, Kundu B, Steffel CN, Varghese T, Meshram NH, Li G, Cook TD, Salamat MS, Dempsey RJ. Transcranial Doppler and Microemboli Detection: Relationships to Symptomatic Status and Histopathology Findings. Ultrasound Med Biol. 2017 Sep;43(9):1861-1867. doi: 10.1016/j.ultrasmedbio.2017.04.025. Epub 2017 Jun 20. PMID 28645797
- [Background] Wang X, Jackson DC, Mitchell CC, Varghese T, Wilbrand SM, Rocque BG, Hermann BP, Dempsey RJ. Classification of Symptomatic and Asymptomatic Patients with and without Cognitive Decline Using Non-invasive Carotid Plaque Strain Indices as Biomarkers. Ultrasound Med Biol. 2016 Apr;42(4):909-18. doi: 10.1016/j.ultrasmedbio.2015.11.025. Epub 2016 Jan 5. PMID 26778288
- [Background] Wang X, Jackson DC, Varghese T, Mitchell CC, Hermann BP, Kliewer MA, Dempsey RJ. Correlation of cognitive function with ultrasound strain indices in carotid plaque. Ultrasound Med Biol. 2014 Jan;40(1):78-89. doi: 10.1016/j.ultrasmedbio.2013.08.001. Epub 2013 Oct 11. PMID 24120415
- [Background] Rocque BG, Jackson D, Varghese T, Hermann B, McCormick M, Kliewer M, Mitchell C, Dempsey RJ. Impaired cognitive function in patients with atherosclerotic carotid stenosis and correlation with ultrasound strain measurements. J Neurol Sci. 2012 Nov 15;322(1-2):20-4. doi: 10.1016/j.jns.2012.05.020. Epub 2012 Jun 1. PMID 22658531
- [Background] McCormick M, Varghese T, Wang X, Mitchell C, Kliewer MA, Dempsey RJ. Methods for robust in vivo strain estimation in the carotid artery. Phys Med Biol. 2012 Nov 21;57(22):7329-53. doi: 10.1088/0031-9155/57/22/7329. Epub 2012 Oct 18. PMID 23079725
- [Background] Dempsey RJ, Vemuganti R, Varghese T, Hermann BP. A review of carotid atherosclerosis and vascular cognitive decline: a new understanding of the keys to symptomology. Neurosurgery. 2010 Aug;67(2):484-93; discussion 493-4. doi: 10.1227/01.NEU.0000371730.11404.36. PMID 20644437
- [Background] Shi H, Varghese T, Dempsey RJ, Salamat MS, Zagzebski JA. Relationship between ultrasonic attenuation, size and axial strain parameters for ex vivo atherosclerotic carotid plaque. Ultrasound Med Biol. 2008 Oct;34(10):1666-77. doi: 10.1016/j.ultrasmedbio.2008.02.014. Epub 2008 May 19. PMID 18490099
- [Background] Wang X, Mitchell CC, Varghese T, Jackson DC, Rocque BG, Hermann BP, Dempsey RJ. Improved Correlation of Strain Indices with Cognitive Dysfunction with Inclusion of Adventitial Layer with Carotid Plaque. Ultrason Imaging. 2016 May;38(3):194-208. doi: 10.1177/0161734615589252. Epub 2015 May 28. PMID 26025578
- [Background] Meshram NH, Varghese T, Mitchell CC, Jackson DC, Wilbrand SM, Hermann BP, Dempsey RJ. Quantification of carotid artery plaque stability with multiple region of interest based ultrasound strain indices and relationship with cognition. Phys Med Biol. 2017 Jul 17;62(15):6341-6360. doi: 10.1088/1361-6560/aa781f. PMID 28594333
- [Background] Barnett PA, Spence JD, Manuck SB, Jennings JR. Psychological stress and the progression of carotid artery disease. J Hypertens. 1997 Jan;15(1):49-55. doi: 10.1097/00004872-199715010-00004. PMID 9050970
- [Background] Pavlovic-Hournac M, Delbauffe D. Protein metabolism in hypo- and hyperstimulated rat thyroid glands. II. Degradation of newly formed thyroidal proteins. Horm Metab Res. 1976 Jan;8(1):55-61. doi: 10.1055/s-0028-1093673. PMID 1248791
- [Background] Nicolaides AN, Kakkos SK, Kyriacou E, Griffin M, Sabetai M, Thomas DJ, Tegos T, Geroulakos G, Labropoulos N, Dore CJ, Morris TP, Naylor R, Abbott AL; Asymptomatic Carotid Stenosis and Risk of Stroke (ACSRS) Study Group. Asymptomatic internal carotid artery stenosis and cerebrovascular risk stratification. J Vasc Surg. 2010 Dec;52(6):1486-1496.e1-5. doi: 10.1016/j.jvs.2010.07.021. PMID 21146746
- [Background] Sztajzel R, Momjian S, Momjian-Mayor I, Murith N, Djebaili K, Boissard G, Comelli M, Pizolatto G. Stratified gray-scale median analysis and color mapping of the carotid plaque: correlation with endarterectomy specimen histology of 28 patients. Stroke. 2005 Apr;36(4):741-5. doi: 10.1161/01.STR.0000157599.10026.ad. Epub 2005 Feb 10. PMID 15705933
- [Background] Mitchell CC, Korcarz CE, Tattersall MC, Gepner AD, Young RL, Post WS, Kaufman JD, McClelland RL, Stein JH. Carotid artery ultrasound texture, cardiovascular risk factors, and subclinical arterial disease: the Multi-Ethnic Study of Atherosclerosis (MESA). Br J Radiol. 2018 Apr;91(1084):20170637. doi: 10.1259/bjr.20170637. Epub 2018 Jan 31. PMID 29308915
- [Background] Welsh KA, Butters N, Mohs RC, Beekly D, Edland S, Fillenbaum G, Heyman A. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part V. A normative study of the neuropsychological battery. Neurology. 1994 Apr;44(4):609-14. doi: 10.1212/wnl.44.4.609. PMID 8164812
- [Background] Fillenbaum GG, van Belle G, Morris JC, Mohs RC, Mirra SS, Davis PC, Tariot PN, Silverman JM, Clark CM, Welsh-Bohmer KA, Heyman A. Consortium to Establish a Registry for Alzheimer's Disease (CERAD): the first twenty years. Alzheimers Dement. 2008 Mar;4(2):96-109. doi: 10.1016/j.jalz.2007.08.005. PMID 18631955
- [Background] Heyman A, Fillenbaum GG, Welsh-Bohmer KA, Gearing M, Mirra SS, Mohs RC, Peterson BL, Pieper CF. Cerebral infarcts in patients with autopsy-proven Alzheimer's disease: CERAD, part XVIII. Consortium to Establish a Registry for Alzheimer's Disease. Neurology. 1998 Jul;51(1):159-62. doi: 10.1212/wnl.51.1.159. PMID 9674796
- [Background] Welsh KA, Fillenbaum G, Wilkinson W, Heyman A, Mohs RC, Stern Y, Harrell L, Edland SD, Beekly D. Neuropsychological test performance in African-American and white patients with Alzheimer's disease. Neurology. 1995 Dec;45(12):2207-11. doi: 10.1212/wnl.45.12.2207. PMID 8848195
- [Background] Fillenbaum GG, Burchett BM, Unverzagt FW, Rexroth DF, Welsh-Bohmer K. Norms for CERAD constructional praxis recall. Clin Neuropsychol. 2011 Nov;25(8):1345-58. doi: 10.1080/13854046.2011.614962. Epub 2011 Oct 13. PMID 21992077
- [Background] Whyte SR, Cullum CM, Hynan LS, Lacritz LH, Rosenberg RN, Weiner MF. Performance of elderly Native Americans and Caucasians on the CERAD Neuropsychological Battery. Alzheimer Dis Assoc Disord. 2005 Apr-Jun;19(2):74-8. doi: 10.1097/01.wad.0000165508.67993.a3. PMID 15942324
- [Background] Ellis G, Rodger J, McAlpine C, Langhorne P. The impact of stroke nurse specialist input on risk factor modification: a randomised controlled trial. Age Ageing. 2005 Jul;34(4):389-92. doi: 10.1093/ageing/afi075. No abstract available. PMID 15955759
- [Background] Vemuganti R. All's well that transcribes well: non-coding RNAs and post-stroke brain damage. Neurochem Int. 2013 Nov;63(5):438-49. doi: 10.1016/j.neuint.2013.07.014. Epub 2013 Aug 15. PMID 23954844
- [Background] Vorlicek J, Mechl Z. [Nephrologic complications of oncologic therapy]. Cas Lek Cesk. 1985 Dec 13;124(50):1561-2. No abstract available. Czech. PMID 4084961
- [Derived] Cress HJ, Mitchell CC, Wilbrand SM, Wesley UV, Morel Valdes GM, Hess T, Varghese T, Maybock J, Metoxen M, Riesenberg A, Vandenberg C, Blohowiak CJ, Kennard J, Danforth D, Dempsey RJ. Methods in Stroke Prevention in the Wisconsin Native American Population. Neuroepidemiology. 2024;58(4):300-309. doi: 10.1159/000536426. Epub 2024 Jan 31. PMID 38295773
- See also: The Oneida Stroke Prevention Program — https://oneidastrokeprogram.wisc.edu/